CLINICAL TRIAL: NCT03248739
Title: A Comparison of External Ventricular Drain Catheter Diameter on Occlusion and Replacement: A Randomized Trial
Brief Title: Comparison of EVD Catheter Diameter on Occlusion and Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Preliminary data did not show a difference. PI decided to terminate study.
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00042079
Record Dates: First submitted 2017-08-04; First posted 2017-08-14 (Actual); Results first posted 2023-10-25 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2022-10

CONDITIONS: Occlusion
Keywords: Catheter; Ventricular; External Ventricular Drain Catheter; EVD Catheter; Occlusion; Ventriculostomy; Clear Bactiseal catheter; Orange Bactiseal catheter; Ventriculostomy Occlusion; Neurosurgery
MeSH Terms: conditions — Bites and Stings

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Clear Bactiseal 'large' catheter (EVD) (Active Comparator): All EVDs will be placed by neurological surgeons in either the major operating suite or in an ICU setting using a previously published protocol. This protocol includes using a burr hole entry point 1 cm anterior to the coronal suture in the mid-pupillary line, prep and sterile drape, pre-procedural antibiotic administration, and tunneling the catheter to an exit site at least 5 cm from the incision. In general, physicians are instructed to first attempt distal irrigation of the drainage chamber using sterile techniques (rarely effective), followed by gentle aspiration of the proximal system and catheter if distal flushing is not effective. If these do not restore patency, a small volume of sterile saline, 3 ml or less, is flushed proximally into the catheter. Patency is checked by lowering the EVD drainage system and evaluating for spontaneous flow through the EVD.
  Interventions: Device: Clear Bactiseal 'large' catheter (EVD)
- Orange Bactiseal 'small' catheter (EVD) (Active Comparator): All EVDs will be placed by neurological surgeons in either the major operating suite or in an ICU setting using a previously published protocol. This protocol includes using a burr hole entry point 1 cm anterior to the coronal suture in the mid-pupillary line, prep and sterile drape, pre-procedural antibiotic administration, and tunneling the catheter to an exit site at least 5 cm from the incision. In general, physicians are instructed to first attempt distal irrigation of the drainage chamber using sterile techniques (rarely effective), followed by gentle aspiration of the proximal system and catheter if distal flushing is not effective. If these do not restore patency, a small volume of sterile saline, 3 ml or less, is flushed proximally into the catheter. Patency is checked by lowering the EVD drainage system and evaluating for spontaneous flow through the EVD.
  Interventions: Device: Orange Bactiseal 'small' catheter (EVD)

INTERVENTIONS:
Device: Clear Bactiseal 'large' catheter (EVD) — Antibiotic-impregnated 'large' catheter (inner diameter 1.9 mm, outer diameter 3.4 mm)
  Arms: Clear Bactiseal 'large' catheter (EVD)
Device: Orange Bactiseal 'small' catheter (EVD) — Antibiotic-impregnated 'small' catheter (inner diameter 1.5 mm, outer diameter 3 mm)
  Arms: Orange Bactiseal 'small' catheter (EVD)

SUMMARY:
A randomized trial comparing small versus large catheters in terms of occlusion and need for replacement to confirm differential occlusion risk based on catheter size. This study will be done to determine whether external ventricular drain catheter diameter has any effect on risk of occlusion.

DETAILED DESCRIPTION:
Ventriculostomy is a common neurosurgical procedure. A Nationwide Inpatient Sample (NIS) database study demonstrated a significant increase in ventriculostomy utilization from 1988-2010, with over 35,000 hospitalizations including a procedural code for ventriculostomy in 2010.

Ventriculostomy occlusion is a common complication after external ventricular drain (EVD) placement. A review of published prospective and retrospective studies indicates that approximately 1-7% of EVDs require replacement secondary to occlusion. Furthermore, in the NIS database study of over 101,000 hospitalizations in which ventriculostomy was performed, nearly 6% of patients required at least one additional ventriculostomy procedure. Studies have demonstrated non-patent EVD in 19-47% of patients, however these studies did not prospectively evaluate EVD occlusion as a primary endpoint, report on number of catheter irrigations performed, or identify risk factors for EVD occlusion.

Recently, the investigators completed a retrospective review of a prospectively collected database of patients undergoing bedside EVD placement with the primary outcome of interest being catheter occlusion. This sample included 101 patients over a 1 year period. Two Codman catheters were available for use (Clear Bactiseal 'large' catheter: outer diameter 3.4 mm, inner diameter 1.9 mm; and Orange Bactiseal 'small' catheter: outer diameter 3 mm, inner diameter 1.5 mm). The decision regarding which catheter to use was made at the time of the procedure based on resident preference and availability. Both temporary occlusion (requiring flushing but patency could be restored) and permanent catheter occlusion (requiring replacement) were common, occurring in 41% and 19% of patients, respectively. Over 25% of small catheters became occluded during the study period compared to 11% of large catheters. Small catheters were associated with a 3.4 times greater odds of occlusion than the larger diameter catheters on multivariable regression analysis. This study suggests that the preferential use of larger diameter catheters may reduce the risk of ventriculostomy occlusion and need for replacement, however the study was not randomized and catheter selection may have been biased.

Recently, a smaller retrospective study of patients with intraventricular hemorrhage performed by Gilard and colleagues demonstrated a lower rate of occlusion and no increased risk of hemorrhage with larger bore catheters. Otherwise, there is no data in the literature supporting the preferential use of catheters based on size (clinical equipoise).

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18-85 years old) with a Glasgow Coma Scale (GCS) score of 7 or higher requiring frontal EVD placement.
* Diagnoses: spontaneous subarachnoid hemorrhage, intraventricular hemorrhage, intraparenchymal or cerebellar hemorrhage due to aneurysm, arteriovenous malformation, arteriovenous fistula, hypertension, or idiopathic etiology.
* Also included are patients for whom the attending neurosurgeon decides that frontal EVD placement is indicated for patient treatment with planned cerebrospinal fluid (CSF) drainage for 72 hours or more.

Exclusion Criteria:

* GCS of 6 or less
* Hunt and Hess subarachnoid hemorrhage grade of 5.
* Age 86 or greater, or age 17 or less.
* Patient cannot consent and next of kin cannot consent prior to procedure.
* Diagnosis of traumatic brain injury, as the EVD is often clamped for extended periods of time.
* Patients anticoagulated prior to admission with warfarin, Effient, Plavix, therapeutic heparin infusion, therapeutic subcutaneous lovenox, therapeutic subcutaneous arixtra, or other therapeutic anticoagulant or antiplatelet agent (ASA not included).
* Plan for EVD placement through non-frontal burr hole.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-06-12 (Actual); Primary Completion 2022-11-04 (Actual); Study Completion 2022-11-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kyle M Fargen, MD, Principal Investigator — Assistant Professor, Surgery Neurosurgery
Locations (1):
- Wake Forest Baptist Health, Winston-Salem, North Carolina, United States

REFERENCES:
- [Background] Rosenbaum BP, Vadera S, Kelly ML, Kshettry VR, Weil RJ. Ventriculostomy: Frequency, length of stay and in-hospital mortality in the United States of America, 1988-2010. J Clin Neurosci. 2014 Apr;21(4):623-32. doi: 10.1016/j.jocn.2013.09.001. PMID 24630243
- [Background] Abla AA, Zabramski JM, Jahnke HK, Fusco D, Nakaji P. Comparison of two antibiotic-impregnated ventricular catheters: a prospective sequential series trial. Neurosurgery. 2011 Feb;68(2):437-42; discussion 442. doi: 10.1227/NEU.0b013e3182039a14. PMID 21135715
- [Background] Tse Ts, Cheng K, Wong K, Pang K, Wong C. Ventriculostomy and Infection: A 4-year-review in a local hospital. Surg Neurol Int. 2010 Sep 9;1:47. doi: 10.4103/2152-7806.69033. PMID 20975968
- [Background] Bauer DF, McGwin G Jr, Melton SM, George RL, Markert JM. The relationship between INR and development of hemorrhage with placement of ventriculostomy. J Trauma. 2011 May;70(5):1112-7. doi: 10.1097/TA.0b013e3181e7c2ae. PMID 20805772
- [Background] Fichtner J, Guresir E, Seifert V, Raabe A. Efficacy of silver-bearing external ventricular drainage catheters: a retrospective analysis. J Neurosurg. 2010 Apr;112(4):840-6. doi: 10.3171/2009.8.JNS091297. PMID 19764827
- [Background] Kakarla UK, Kim LJ, Chang SW, Theodore N, Spetzler RF. Safety and accuracy of bedside external ventricular drain placement. Neurosurgery. 2008 Jul;63(1 Suppl 1):ONS162-6; discussion ONS166-7. doi: 10.1227/01.neu.0000335031.23521.d0. PMID 18728595
- [Background] Khanna RK, Rosenblum ML, Rock JP, Malik GM. Prolonged external ventricular drainage with percutaneous long-tunnel ventriculostomies. J Neurosurg. 1995 Nov;83(5):791-4. doi: 10.3171/jns.1995.83.5.0791. PMID 7472544
- [Background] Bogdahn U, Lau W, Hassel W, Gunreben G, Mertens HG, Brawanski A. Continuous-pressure controlled, external ventricular drainage for treatment of acute hydrocephalus--evaluation of risk factors. Neurosurgery. 1992 Nov;31(5):898-903; discussion 903-4. doi: 10.1227/00006123-199211000-00011. PMID 1436414
- [Background] Olson DM, Zomorodi M, Britz GW, Zomorodi AR, Amato A, Graffagnino C. Continuous cerebral spinal fluid drainage associated with complications in patients admitted with subarachnoid hemorrhage. J Neurosurg. 2013 Oct;119(4):974-80. doi: 10.3171/2013.6.JNS122403. Epub 2013 Aug 20. PMID 23957382
- [Background] Chi H, Chang KY, Chang HC, Chiu NC, Huang FY. Infections associated with indwelling ventriculostomy catheters in a teaching hospital. Int J Infect Dis. 2010 Mar;14(3):e216-9. doi: 10.1016/j.ijid.2009.04.006. Epub 2009 Jul 31. PMID 19647466
- [Background] Gilard V, Djoubairou BO, Lepetit A, Metayer T, Gakuba C, Gourio C, Derey S, Proust F, Emery E, Gaberel T. Small versus Large Catheters for Ventriculostomy in the Management of Intraventricular Hemorrhage. World Neurosurg. 2017 Jan;97:117-122. doi: 10.1016/j.wneu.2016.09.105. Epub 2016 Oct 10. PMID 27729301
- [Background] Rahman M, Whiting JH, Fauerbach LL, Archibald L, Friedman WA. Reducing ventriculostomy-related infections to near zero: the eliminating ventriculostomy infection study. Jt Comm J Qual Patient Saf. 2012 Oct;38(10):459-64. doi: 10.1016/s1553-7250(12)38061-6. PMID 23130392

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 33 subjects were consented to study with 33 being randomized.
Groups:
- Large Bore Catheter Group: Large Bore Catheter (1.9mmID)
- Small Bore Catheter Group: Small Bore Catheter (1.5mm ID)
Period: Overall Study
Arm/Group | Large Bore Catheter Group | Small Bore Catheter Group
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Large: Large Bore Catheter (1.9mmID)
- Small: Small Bore Catheter (1.5mm ID)
- Total: Total of all reporting groups
Arm/Group | Large | Small | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.8 (13.9) | 62.1 (13.1) | 60.5 (13.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 9 | 19
  Male | 7 | 7 | 14
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 17 | 16 | 33
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 3 | 3 | 6
  White | 13 | 13 | 26
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Permanent Catheter Occlusions
Description: This is defined by a non-functioning (non-patent) EVD where patency cannot be restored through catheter manipulation or flushing.
Time Frame: Up to 4 weeks
Population: Randomized to Large or Small Bore Catheters
Measure: Count of Participants; unit: Participants
Arm/Group | Large | Small
Number analyzed (Participants) | 17 | 16
Participants | 0 | 2
Statistical Analysis 1: Comparison: Large vs Small; Test type: Equivalence — Based on occlusion data from the previously referenced prospective study, as well as a P-value of 0.05 and power of 0.80, the study will need to include 90 patients to demonstrate statistical significance. To ensure that power is adequate, we will plan to enroll 120 patients (60 in each arm); p = 0.23, Fisher Exact

2. Secondary Outcome: Number of Participants With Catheter Replacements
Description: Defined by replacement of the ipsilateral EVD due to permanent occlusion, or placement of a contralateral EVD in the setting of a non-functioning ipsilateral catheter. Catheters placed contralaterally in the setting of a functioning ipsilateral catheter will not be considered replacements.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Large | Small
Number analyzed (Participants) | 17 | 16
Participants | 1 | 3

3. Secondary Outcome: Number of Participants With Temporary Occlusions
Description: Defined by non-functioning (non-patent) catheter requiring neurosurgeon flushing or manipulation in order to restore patency. By definition, such maneuvers must restore patency of the EVD such that it is functioning normally afterwards. Multiple temporary occlusions may be possible.
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Large | Small
Number analyzed (Participants) | 17 | 16
Participants | 2 | 0

4. Secondary Outcome: Number of Participants With Procedure-related Hemorrhages
Description: Presence of new catheter-related intraparenchymal hemorrhage, subdural hematoma, or intraventricular hemorrhage on CT scan 48 hours after placement.
Time Frame: 48 hours after placement.
Measure: Count of Participants; unit: Participants
Arm/Group | Large | Small
Number analyzed (Participants) | 17 | 16
Participants | 0 | 0

5. Secondary Outcome: Number of Participants With Symptomatic Hemorrhages
Description: Presence of new neurologic deficits as a result of EVD-related hemorrhage, or resulting in need for further procedures due to new EVD-related hemorrhage (craniotomy for hematoma evacuation, ICP monitoring, etc).
Time Frame: Up to 4 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Large | Small
Number analyzed (Participants) | 17 | 16
Participants | 0 | 0

ADVERSE EVENTS:
Time Frame: 4 weeks
Arm/Group | Large | Small
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol (2019-11-03): https://cdn.clinicaltrials.gov/large-docs/39/NCT03248739/Prot_001.pdf
  • Informed Consent Form (2022-09-12): https://cdn.clinicaltrials.gov/large-docs/39/NCT03248739/ICF_000.pdf